CLINICAL TRIAL: NCT03549078
Title: A Randomized Evaluation of a Multidimensional Behavioral Intervention for Those at Risk for Alzheimer's Dementia
Brief Title: A Multidimensional Behavioral Intervention for Those at Risk for Alzheimer's Dementia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Davis (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 967764
Record Dates: First submitted 2018-05-15; First posted 2018-06-07 (Actual); Last update posted 2020-06-11 (Actual); Status verified 2020-06

CONDITIONS: Functional Aging; Subjective Cognitive Concerns; Compensation Strategies; Brain Health Activities
MeSH Terms: interventions — Methods

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention (Experimental): Participants will complete an initial assessment within 2 weeks prior to starting the course or during the first class. The course will include 10 sessions conducted on a weekly basis. Following completion of the course, participants will again complete another assessment during the last class or within 2 weeks of course completion. Participants may be invited to complete assessments at 3- and 6-months following course completion.
  Interventions: Behavioral: Intervention

INTERVENTIONS:
Behavioral: Intervention — Subjects will attend a series of 2 hour classes, once a week for 10 weeks. Topics discussed in group sessions will cover compensation strategies (e.g., calendar, goal setting and task lists, functional zones) and brain health behaviors (e.g., exercise, cognitive activity, stress reduction and mindfulness).
  Subjects may be asked to wear an actigraphy monitor (that looks like a wrist watch) and/or heart rate sensor that is designed to collect information regarding physical activity.

SUMMARY:
This intervention is designed to promote enhanced use of compensation strategies including calendar and task list use, and organization systems, as well as increased engagement with brain health activities including physical exercise, cognitive activities, and stress reduction.

DETAILED DESCRIPTION:
The purpose of this study is to test the feasibility and efficacy of a 10-week multi-dimensional intervention for older adults with subjective cognitive concerns (SCC). The goal of this intervention is to enhance compensation skills related to everyday executive and everyday memory functions through training in the systematic use of a calendar system, goal setting and task list system, and organizational strategies within the context of the individual's daily life. This multidimensional intervention program also targets engagement in healthy lifestyle activities (physical exercise, intellectual stimulation, positive emotional functioning) to further promote brain health and functional resilience. Importantly, both treatment components work synergistically as the use of compensation strategies assists in building healthy activities into daily routines (e.g., scheduling exercise into one's calendar and putting it on a task list).

ELIGIBILITY:
Inclusion Criteria:

* A positive complaint in response to two questions ('Do you feel like your memory or other aspects of thinking are becoming worse?'; 'Does this worry you?')
* normal cognitive performance corrected for age and education on a global measure of cognitive functioning
* independent in all activities of daily living.
* English speaking;
* Available informant to complete surveys;
* Ambulatory

Exclusion Criteria:

* Known neurological condition;
* Severe psychiatric illness (e.g., current depression).

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 69 (Actual)
Dates: Start 2017-01-01 (Actual); Primary Completion 2019-08-14 (Actual); Study Completion 2019-08-14 (Actual)

PRIMARY OUTCOMES:
Everyday Compensation Questionnaire | Change from baseline to immediately post-intervention and through 6 month follow up
  a 54-item self-report questionnaire that asks participants how often they engage in a variety of activities that help them stay cognitively and physically active.
Everyday Cognition | Change from baseline to immediately post-intervention and through 6 month follow up
  self-rated questionnaire of cognitively-based everyday abilities. The ECog comprises of 39 items on which the participant's current level of everyday functioning is compared to 10 years earlier. Items are rated on a four-point scale: 1= better or no change compared to 10 years earlier; 4= consistently much worse. Higher scores indicate greater functional limitations

SECONDARY OUTCOMES:
Beck Depression Inventory | Measured at baseline, immediately after intervention, and 3 and 6 month follow up visits
  Measures depressive symptomatology
Beck Anxiety Inventory | Measured at baseline, immediately after intervention, and 3 and 6 month follow up visits
  Measures anxiety symptomatology
List learning task | Measured at baseline, immediately after intervention, and 3 and 6 month follow up visits
  measures learning and memory
Executive function task | Measured at baseline, immediately after intervention, and 3 and 6 month follow up visits
  measures executive function
psychomotor speed task | Measured at baseline, immediately after intervention, and 3 and 6 month follow up visits
  measures psychomotor speed function
GRIT | Measured at baseline, immediately after intervention, and 3 and 6 month follow up visits
  an 8-item questionnaire assessing consistency of interest and perseverance of effort on a five-point scale: 1 = not at all like me, 5 = very much like me.

CONTACTS AND LOCATIONS:
Overall Officials: Katherine G Denny, PhD, Principal Investigator — University of California, Davis
Locations (1):
- University of California Davis, Sacramento, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Tomaszewski Farias S, Schmitter-Edgecombe M, Weakley A, Harvey D, Denny KG, Barba C, Gravano JT, Giovannetti T, Willis S. Compensation Strategies in Older Adults: Association With Cognition and Everyday Function. Am J Alzheimers Dis Other Demen. 2018 May;33(3):184-191. doi: 10.1177/1533317517753361. Epub 2018 Jan 23. PMID 29357670
- [Background] Farias ST, Lau K, Harvey D, Denny KG, Barba C, Mefford AN. Early Functional Limitations in Cognitively Normal Older Adults Predict Diagnostic Conversion to Mild Cognitive Impairment. J Am Geriatr Soc. 2017 Jun;65(6):1152-1158. doi: 10.1111/jgs.14835. Epub 2017 Mar 17. PMID 28306147
- [Background] Greenaway MC, Duncan NL, Smith GE. The memory support system for mild cognitive impairment: randomized trial of a cognitive rehabilitation intervention. Int J Geriatr Psychiatry. 2013 Apr;28(4):402-9. doi: 10.1002/gps.3838. Epub 2012 Jun 7. PMID 22678947
- [Background] Greenaway MC, Hanna SM, Lepore SW, Smith GE. A behavioral rehabilitation intervention for amnestic mild cognitive impairment. Am J Alzheimers Dis Other Demen. 2008 Oct-Nov;23(5):451-61. doi: 10.1177/1533317508320352. PMID 18955724
- [Background] Lau KM, Parikh M, Harvey DJ, Huang CJ, Farias ST. Early Cognitively Based Functional Limitations Predict Loss of Independence in Instrumental Activities of Daily Living in Older Adults. J Int Neuropsychol Soc. 2015 Oct;21(9):688-98. doi: 10.1017/S1355617715000818. Epub 2015 Sep 22. PMID 26391766
- [Derived] Denny KG, Chan ML, Gravano J, Harvey D, Meyer OL, Huss O, Farias ST. A randomized control trial of a behavioral intervention for older adults with subjective cognitive complaints that combines cognitive rehabilitation strategies and lifestyle modifications. Neuropsychol Dev Cogn B Aging Neuropsychol Cogn. 2023 Jan;30(1):78-93. doi: 10.1080/13825585.2021.1965530. Epub 2021 Aug 19. PMID 34412558